CLINICAL TRIAL: NCT07084493
Title: *Effect of Prophylactic Common Bile Duct Stenting Versus Non Stenting on Recurrence of Common Bile Duct Stones in Patients Awaiting Cholecystectomy*
Brief Title: *Effect of Prophylactic CBD Stenting Versus Non Stenting on Recurrence of CBD Stones in Patients Awaiting Cholecystectomy*
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Huda Mokhtar Salim, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ERCP in CBD stones
Record Dates: First submitted 2025-07-15; First posted 2025-07-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Calcular Obstructive Jaundice
Keywords: CBD stones, ERCP

STUDY DESIGN:
Intervention Model Description: Following ERCP and biliary duct clearance, participants will be randomly assigned in a 1:1 ratio to either:
  Stent Group: Placement of a prophylactic CBD stent will be placed. Control Group: No stent placement after biliary clearance. Patients will be monitored every month until cholecystectomy or up to 3 months, whichever comes first.
  Follow-up includes:
  Clinical assessment. LFTs and pancreatic enzymes. Imaging: US (MRCP if symptomatic). Stent removal (if placed) at 3 months or earlier if symptomatic. Repeat ERCP for recurrence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CASE WITH cbd STONES (Active Comparator): Age > 18 years.
  Documented CBD stones by various imaging or ERCP.
  Successful biliary clearance by ERCP.
  Scheduled for elective cholecystectomy within 3 months.
  Provide written informed consent.
  Interventions: Device: CBD stent either a 7-Fr and 7 cm or a 10-Fr and 7-cm OR double-pigtail stent; Device: biliary stent

INTERVENTIONS:
Device: CBD stent either a 7-Fr and 7 cm or a 10-Fr and 7-cm OR double-pigtail stent — prophylactic CBD stent either a 7-Fr and 7 cm or a 10-Fr and 7-cm double-pigtail stent
Device: biliary stent — prophylactic CBD stent either a 7-Fr and 7 cm or a 10-Fr and 7-cm double-pigtail stent

SUMMARY:
Primary objective:

Compare recurrence rates of CBD stones in stented versus non-stented patients.

Secondary objectives:

Identify predictors of stone recurrence. Assess the incidence and risk factors for post-ERCP complications. Evaluate time to recurrence and rate of hospital readmissions. Explore impact on quality of life and ease of subsequent cholecystectomy.

DETAILED DESCRIPTION:
Choledocholithiasis, the presence of stones in the common bile duct (CBD), occurs in 10-20% of patients with symptomatic gallstones and can lead to severe complications such as obstructive jaundice, cholangitis, and pancreatitis Endoscopic retrograde cholangiopancreatography (**ERCP**) with stone extraction is the gold standard treatment, achieving >90% success rates in ductal clearance.

Despite successful initial clearance, CBD stone recurrence remains a significant issue, with reported rates ranging from 4% to 24% .

To reduce recurrence, prophylactic biliary stenting has been proposed, particularly in high-risk patients (e.g., large or multiple stones, dilated CBD, periampullary diverticulum) However, its routine use remains controversial due to conflicting evidence on efficacy, stent-related complications (e.g., migration, occlusion, cholangitis), and increased healthcare costs.

ELIGIBILITY:
"Inclusion Criteria":

* Age > 18 years.
* Documented CBD stones by various imaging or ERCP.
* Successful biliary clearance by ERCP.
* Scheduled for elective cholecystectomy within 3 months.
* Provide written informed consent.

"Exclusion Criteria":

* Previous biliary surgery.
* Known malignancy involving the biliary system.
* Comorbid conditions preventing surgery such as bleeding tendency.
* Pregnancy.
* Failure to obtain consent.
* Failed stone clearance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of CBD stones within 3 months, confirmed by imaging or ERCP. | 3 months
  Recurrence of CBD stones within 3 months, confirmed by imaging or ERCP.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
SPSS version 22 will be used. Continuous variables: mean ± SD or median (IQR), compared via t-test or Mann-Whitney.
  Categorical variables: chi-square or Fisher's exact test. Kaplan-Meier for time-to-event outcomes. Multivariate regression to identify predictors. P < 0.05 considered significant.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/26343220